CLINICAL TRIAL: NCT02457793
Title: A Phase Ib, Open-Label, Dose-Escalation Study Of The Safety, Tolerability, and Pharmacokinetics of Cobimetinib and GDC-0994 In Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of the Safety, Tolerability, and Effects of Cobimetinib and GDC-0994 in Patients With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO29653; 2015-000092-27 (EudraCT Number)
Record Dates: First submitted 2015-05-27; First posted 2015-05-29 (Estimated); Results first posted 2018-08-24 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Non-Small Cell Lung Cancer, Metastatic Colorectal Cancer, Metastatic Non Small Cell Lung Cancer, Metastatic Cancers, Melanoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Neoplasms; Melanoma | interventions — cobimetinib; ravoxertinib

ARMS (6):
- Not assigned (Experimental): One participant was assigned to receive intermittent cobimetinib 80 milligrams (mg) + GDC 0994 200 mg) and did receive study drug. However, the participant diary was not returned, and the site was unable to document study dose administration.
  Interventions: Drug: Cobimetinib; Drug: GDC-0994
- COB 20 mg + GDC 200 mg (Experimental): Concurrent or intermittent dosing of cobimetinib 20 mg, concurrent with GDC-0994 200 mg for 21 consecutive days, followed by 7 days off.
  Interventions: Drug: Cobimetinib; Drug: GDC-0994
- COB 40 mg + GDC 200 mg (Experimental): Concurrent or intermittent dosing of cobimetinib 40 mg, concurrent with GDC-0994 200 mg for 21 consecutive days, followed by 7 days off.
  Interventions: Drug: Cobimetinib; Drug: GDC-0994
- COB 80 mg + GDC 200 mg (Experimental): Concurrent or intermittent dosing of cobimetinib 80 mg, concurrent with GDC-0994 200 mg for 21 consecutive days, followed by 7 days off.
  Interventions: Drug: Cobimetinib; Drug: GDC-0994
- COB 80 mg + GDC 400 mg (Experimental): Concurrent or intermittent dosing of cobimetinib 80 mg, concurrent with GDC-0994 400 mg for 21 consecutive days, followed by 7 days off.
  Interventions: Drug: Cobimetinib; Drug: GDC-0994
- COB 100 mg + GDC 200 mg (Experimental): Concurrent or intermittent dosing of cobimetinib 100 mg, concurrent with GDC-0994 200 mg for 21 consecutive days, followed by 7 days off.
  Interventions: Drug: Cobimetinib; Drug: GDC-0994

INTERVENTIONS:
Drug: Cobimetinib — Cobimetinib given concurrently or intermittently with GDC-0994 for 21 consecutive days followed by 7 days off.
Drug: GDC-0994 — GDC-0994 given for 21 consecutive days followed by 7 days off, along with concurrent or intermittent dosing of cobimetinib.

SUMMARY:
This is a two-stage dose-escalation study to assess the safety, tolerability and effects of oral dosing of cobimetinib and GDC-0994 administered in combination in patients with histologically confirmed, locally advanced, or metastatic solid tumors for which standard therapies either do not exist or have proven ineffective or intolerable.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Histologically or cytologically documented, locally advanced or metastatic solid tumors for which standard therapy either does not exist or has proven ineffective or intolerable
* Evaluable disease or disease measurable
* Life expectancy > or = 12 weeks
* Adequate hematologic and end organ function
* For female patients of childbearing potential and male patients with partners of childbearing potential, use of an effective form of contraception with continued use for study duration and up to 3 months or more following discontinuation of treatment drug
* Fluorodeoxyglucose positron emission tomography (FDG-PET) avid disease on baseline scan

For enrollment in part 2, patients must meet all of the following:

* Measurable disease
* No more than four prior systemic therapies for locally advanced or metastatic cancer

Exclusion Criteria:

* History of prior significant toxicity from another MEK inhibitor or ERK inhibitor requiring discontinuation of treatment
* Evidence of visible retinal pathology as assessed by ophthalmologic examination that is considered a risk factor for retinal vein thrombosis
* History of glaucoma
* Intraocular pressure > 21 mmHg as measured by tonometry
* Predisposing factors to retinal vein occlusion (RVO)
* History of RVO, neurosensory retinal detachment, or neovascular macular degeneration
* Allergy or hypersensitivity to components of the cobimetinib or GDC-0994 formulation
* Palliative radiotherapy within 2 weeks prior to first dose of study-drug treatment in Cycle 1
* Experimental therapy within 4 weeks prior to first dose of study-drug treatment in Cycle 1
* Major surgical procedure or significant traumatic injury within 4 weeks prior to the first dose of study-drug treatment in Cycle 1, or anticipation of the need for major surgery during the course of study treatment
* Anti-cancer therapy within 28 days prior to the first dose of study-drug treatment in Cycle 1
* Current severe, uncontrolled systemic disease
* History of clinically significant cardiac dysfunction
* History of symptomatic congestive heart failure or serious cardiac arrhythmia requiring treatment
* History of myocardial infarction within 6 months prior to the first dose of study-drug treatment in Cycle 1
* History of congenital long QT syndrome or QTc > 470 msec
* LVEF
* History of malabsorption or other condition that would interfere with enteral absorption
* Clinically significant history of liver disease, current alcohol abuse, or current known active infection with HIV, hepatitis B virus, or hepatitis C virus
* Any condition requiring warfarin or thrombolytic anticoagulants
* Active autoimmune disease
* Uncontrolled ascites requiring weekly large volume paracentesis for 3 consecutive weeks prior to enrollment
* Pregnancy, lactation, or breastfeeding
* Known brain metastases that are untreated, symptomatic, or require therapy to control symptoms
* No other history of or ongoing malignancy that would potentially interfere with the interpretation of the Pharmacodynamic (PD) or efficacy assays

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-06-16 (Actual); Primary Completion 2016-12-05 (Actual); Study Completion 2016-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (5):
- United States (5):
  - University of Colorado, Aurora, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Sarah Cannon Research Institute, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Not Assigned | COB 20 mg + GDC 200 mg | COB 40 mg + GDC 200 mg | COB 80 mg + GDC 200 mg | COB 80 mg + GDC 400 mg | COB 100 mg + GDC 200 mg
Started | 1 | 5 | 3 | 5 | 4 | 6
Completed | 0 | 1 | 0 | 0 | 0 | 0
Not Completed | 1 | 4 | 3 | 5 | 4 | 6
Not completed — Reason not specified | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 4 | 2 | 2 | 2 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 1 | 1 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Not Assigned | COB 20 mg + GDC 200 mg | COB 40 mg + GDC 200 mg | COB 80 mg + GDC 200 mg | COB 80 mg + GDC 400 mg | COB 100 mg + GDC 200 mg | Total
Number analyzed (Participants) | 1 | 5 | 3 | 5 | 4 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.0 (9999) | 53.0 (11.5) | 57.3 (11.0) | 51.6 (14.2) | 52.3 (5.6) | 59.7 (11.5) | 54.6 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 5 | 3 | 4 | 2 | 3 | 17
  Male | 1 | 0 | 0 | 1 | 2 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLTs)
Description: DLTs include symptoms considered by the investigator to be possibly related to study drug.
Time Frame: 28 days (Cycle 1)
Population: All participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Not Assigned | COB 20 mg + GDC 200 mg | COB 40 mg + GDC 200 mg | COB 80 mg + GDC 200 mg | COB 80 mg + GDC 400 mg | COB 100 mg + GDC 200 mg
Number analyzed (Participants) | 1 | 5 | 3 | 5 | 4 | 6
Participants
  Dermatitis Acneiform | 1 | 0 | 0 | 0 | 0 | 0
  Rash | 1 | 0 | 0 | 0 | 0 | 0
  Diarrhoea | 0 | 0 | 1 | 0 | 0 | 0
  Myocardial infarction | 0 | 0 | 0 | 1 | 0 | 0

2. Primary Outcome: Percentage of Participants With at Least One Adverse Event
Description: An adverse event is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of causal attribution.
Time Frame: Up to 15 months
Population: All participants.
Measure: Number; unit: percentage of participants
Arm/Group | Not Assigned | COB 20 mg + GDC 200 mg | COB 40 mg + GDC 200 mg | COB 80 mg + GDC 200 mg | COB 80 mg + GDC 400 mg | COB 100 mg + GDC 200 mg
Number analyzed (Participants) | 1 | 5 | 3 | 5 | 4 | 6
percentage of participants | 100 | 100 | 100 | 100 | 100 | 100

3. Primary Outcome: Percentage of Participants With at Least One Adverse Event of Special Interest
Description: AESIs were graded per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), v4.0. AESIs included the following: Grade ≥ 1 retinal vein occlusion; Grade ≥ 2 visual disturbances (including events suggestive of serous retinopathy); Grade ≥ 3 rash for > 7 days; Grade ≥ 3 diarrhea for > 3 days; Grade ≥ 2 left ventricular ejection fraction (LVEF) decrease; Grade 3 hepatotoxicity; any dose-limiting toxicity (DLT); cases of potential drug-induced liver injury that include an elevated alanine aminotransferase (ALT) or aspartate aminotransferase (AST) (AST > 3 × baseline value [and above the upper limit of normal, ULN]) in combination with either an elevated bilirubin ( > 2 × ULN) or clinical jaundice; or suspected transmission of an infectious agent by either study drug.
Time Frame: Up to 15 months
Population: All participants.
Measure: Number; unit: percentage of participants
Arm/Group | Not Assigned | COB 20 mg + GDC 200 mg | COB 40 mg + GDC 200 mg | COB 80 mg + GDC 200 mg | COB 80 mg + GDC 400 mg | COB 100 mg + GDC 200 mg
Number analyzed (Participants) | 1 | 5 | 3 | 5 | 4 | 6
percentage of participants | 100.0 | 100 | 33.3 | 60.0 | 75.0 | 50.0

4. Primary Outcome: Percentage of Participants With at Least One Serious Adverse Event (SAE)
Description: A SAE is any experience that: results in death, is life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is medically significant.
Time Frame: Up to 15 months
Population: All participants.
Measure: Number; unit: percentage of participants
Arm/Group | Not Assigned | COB 20 mg + GDC 200 mg | COB 40 mg + GDC 200 mg | COB 80 mg + GDC 200 mg | COB 80 mg + GDC 400 mg | COB 100 mg + GDC 200 mg
Number analyzed (Participants) | 1 | 5 | 3 | 5 | 4 | 6
percentage of participants | 100.0 | 40.0 | 66.7 | 60.0 | 50.0 | 66.7

5. Primary Outcome: Percentage of Participants With Laboratory Abnormalities
Description: Laboratory abnormalities were graded per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), v4.0.
  SGPT/ALT - serum glutamic-pyruvic transaminase/alanine aminotransferase; SGOT/AST - serum glutamic oxaloacetic transaminase/aspartate aminotransferase
Time Frame: Up to 15 months
Population: All participants. Data are reported for evaluable participants.
Measure: Number; unit: percentage of participants
Arm/Group | Not Assigned | COB 20 mg + GDC 200 mg | COB 40 mg + GDC 200 mg | COB 80 mg + GDC 200 mg | COB 80 mg + GDC 400 mg | COB 100 mg + GDC 200 mg
Number analyzed (Participants) | 1 | 5 | 3 | 5 | 4 | 6
percentage of participants
  Albumin | 100.0 | 80.0 | 66.7 | 100.0 | 100.0 | 83.3
  Alkaline Phosphatase | 100.0 | 80.0 | 66.7 | 80.0 | 75.0 | 50.0
  SGPT/ALT | 0.0 | 60.0 | 0.0 | 60.0 | 25.0 | 33.3
  SGOT/AST | 100.0 | 100.0 | 66.7 | 60.0 | 75.0 | 50.0
  Calcium | 100.0 | 20.0 | 33.3 | 80.0 | 100.0 | 33.3
  Creatinine | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 50.0
  Blood Glucose, Fasting: number analyzed (Participants) | 1 | 4 | 2 | 3 | 3 | 1
  Blood Glucose, Fasting | 0.0 | 100.0 | 100.0 | 0.0 | 66.6 | 100.0
  Gamma Glutamyl Transferase | 100.0 | 60.0 | 66.7 | 60.0 | 75.0 | 50.0
  Glucose: number analyzed (Participants) | 1 | 5 | 3 | 5 | 3 | 6
  Glucose | 0 | 20.0 | 0.0 | 0.0 | 0.0 | 0.0
  Hemoglobin | 100.0 | 60.0 | 66.7 | 100.0 | 75.0 | 66.7
  Lymphocytes, Absolute | 100.0 | 40.0 | 33.3 | 60.0 | 50.0 | 16.7
  Magnesium | 100.0 | 40.0 | 66.6 | 20.0 | 50.0 | 16.7
  Phosphorus | 0.0 | 20.0 | 0.0 | 0.0 | 25.0 | 0.0
  Platelets | 0.0 | 20.0 | 33.3 | 40.0 | 50.0 | 33.3
  Potassium | 0.0 | 40.0 | 66.7 | 40.0 | 25.0 | 33.3
  Sodium | 0.0 | 60.0 | 33.3 | 0.0 | 50.0 | 16.7
  Bilirubin | 100.0 | 20.0 | 0.0 | 0.0 | 25.0 | 0.0
  Uric Acid | 0.0 | 20.0 | 0.0 | 0.0 | 25.0 | 16.7
  White Blood Cell Count | 0.0 | 20 | 0.0 | 20.0 | 25.0 | 33.3

6. Primary Outcome: Mean Change From Baseline in Diastolic Blood Pressure
Time Frame: Baseline, up to 15 months
Population: All participants. Data are reported for evaluable participants.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Not Assigned | COB 20 mg + GDC 200 mg | COB 40 mg + GDC 200 mg | COB 80 mg + GDC 200 mg | COB 80 mg + GDC 400 mg | COB 100 mg + GDC 200 mg
Number analyzed (Participants) | 0 | 5 | 3 | 2 | 1 | 5
millimeters of mercury (mmHg) |  | -4.2 (7.6) | -4.3 (11.8) | -0.5 (7.8) | 29.0 | -13.2 (15.9)

7. Primary Outcome: Mean Change From Baseline in Lean Body Mass
Time Frame: Baseline, Day 15
Population: All participants. Data are reported for evaluable participants.
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Not Assigned | COB 20 mg + GDC 200 mg | COB 40 mg + GDC 200 mg | COB 80 mg + GDC 200 mg | COB 80 mg + GDC 400 mg | COB 100 mg + GDC 200 mg
Number analyzed (Participants) | 0 | 4 | 1 | 5 | 3 | 2
kilograms (kg) |  | 0.25 (1.26) | -2.00 | -0.20 (1.30) | -4.33 (5.77) | 0.00 (1.41)

8. Primary Outcome: Mean Change From Baseline in Pulse Rate
Time Frame: Baseline, up to 15 months
Population: All participants. Data are reported for evaluable participants.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Not Assigned | COB 20 mg + GDC 200 mg | COB 40 mg + GDC 200 mg | COB 80 mg + GDC 200 mg | COB 80 mg + GDC 400 mg | COB 100 mg + GDC 200 mg
Number analyzed (Participants) | 0 | 5 | 3 | 2 | 1 | 5
beats per minute |  | 20.4 (32.7) | 16.7 (22.7) | 15.5 (9.2) | 43.0 | 12.2 (21.6)

9. Primary Outcome: Mean Change From Baseline in Respiratory Rate
Time Frame: Baseline, up to 15 months
Population: All participants. Data are reported for evaluable participants.
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Not Assigned | COB 20 mg + GDC 200 mg | COB 40 mg + GDC 200 mg | COB 80 mg + GDC 200 mg | COB 80 mg + GDC 400 mg | COB 100 mg + GDC 200 mg
Number analyzed (Participants) | 0 | 5 | 3 | 2 | 1 | 5
breaths per minute |  | 1.6 (3.6) | 0.3 (0.6) | 0.0 (0.0) | 2.0 | 1.6 (3.6)

10. Primary Outcome: Mean Change From Baseline in Systolic Blood Pressure
Time Frame: Baseline, up to 15 months
Population: All participants. Data are reported for evaluable participants.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Not Assigned | COB 20 mg + GDC 200 mg | COB 40 mg + GDC 200 mg | COB 80 mg + GDC 200 mg | COB 80 mg + GDC 400 mg | COB 100 mg + GDC 200 mg
Number analyzed (Participants) | 0 | 5 | 3 | 2 | 1 | 5
mmHg |  | 2.2 (19.6) | -4.0 (30.6) | -1.5 (0.7) | 34.0 | -17.2 (20.9)

11. Primary Outcome: Mean Change From Baseline in Temperature
Time Frame: Baseline, up to 15 months
Population: All participants. Data are reported for evaluable participants.
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Not Assigned | COB 20 mg + GDC 200 mg | COB 40 mg + GDC 200 mg | COB 80 mg + GDC 200 mg | COB 80 mg + GDC 400 mg | COB 100 mg + GDC 200 mg
Number analyzed (Participants) | 0 | 5 | 3 | 2 | 1 | 5
degrees Celsius |  | -0.04 (0.31) | -0.20 (0.87) | -0.16 (0.20) | -0.20 | -0.16 (0.34)

12. Primary Outcome: Mean Change From Baseline in Weight
Time Frame: Baseline, up to 15 months
Population: All participants. Data are reported for evaluable participants.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Not Assigned | COB 20 mg + GDC 200 mg | COB 40 mg + GDC 200 mg | COB 80 mg + GDC 200 mg | COB 80 mg + GDC 400 mg | COB 100 mg + GDC 200 mg
Number analyzed (Participants) | 0 | 5 | 3 | 2 | 1 | 5
kg |  | -4.01 (7.71) | 0.33 (1.69) | 0.57 (3.34) | -2.70 | -0.80 (3.43)

13. Secondary Outcome: Maximum Serum Concentration (Cmax) for GDC-0994
Time Frame: Up to Day 22
Population: Data are reported for evaluable participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micromoles
Groups:
- COB 80 mg + GDC 300 mg: Concurrent or intermittent dosing of cobimetinib 80 mg, concurrent with GDC-0994 300 mg for 21 consecutive days, followed by 7 days off.
Arm/Group | COB 80 mg + GDC 300 mg | COB 20 mg + GDC 200 mg | COB 40 mg + GDC 200 mg | COB 80 mg + GDC 200 mg | COB 80 mg + GDC 400 mg | COB 100 mg + GDC 200 mg
Number analyzed (Participants) | 1 | 5 | 3 | 5 | 4 | 6
micromoles
  Day 1: number analyzed (Participants) | 0 | 5 | 3 | 5 | 4 | 6
  Day 1 |  | 2.51 (54.6) | 2.08 (68.4) | 2.02 (109.0) | 2.42 (33.6) | 2.56 (77.8)
  Steady State: number analyzed (Participants) | 1 | 2 | 1 | 3 | 1 | 2
  Steady State | 2.56 | 1.80 (74.2) | 2.01 (0.0) | 2.26 (23.1) | 2.09 (0.0) | 2.36 (28.2)

14. Secondary Outcome: Median Time to Maximum Serum Concentration (Tmax) for GDC-0994
Time Frame: Up to Day 22
Population: Data are reported for evaluable participants.
Measure: Mean (Full Range); unit: hours
Arm/Group | COB 80 mg + GDC 300 mg | COB 20 mg + GDC 200 mg | COB 40 mg + GDC 200 mg | COB 80 mg + GDC 200 mg | COB 80 mg + GDC 400 mg | COB 100 mg + GDC 200 mg
Number analyzed (Participants) | 1 | 5 | 3 | 5 | 4 | 6
hours
  Day 1: number analyzed (Participants) | 0 | 5 | 3 | 5 | 4 | 6
  Day 1 |  | 4.00 [2.00 to 6.00] | 6.00 [2.00 to 6.00] | 3.00 [2.00 to 24.0] | 15.0 [2.0 to 24.0] | 2.50 [1.00 to 4.00]
  Steady State: number analyzed (Participants) | 1 | 2 | 1 | 3 | 1 | 2
  Steady State | 3.00 | 3.00 [2.00 to 4.00] | 24.0 | 2.00 [2.00 to 3.00] | 3.00 | 2.00 [2.00 to 2.00]

15. Secondary Outcome: Maximum Serum Concentration (Cmax) for Cobimetinib
Time Frame: Up to Day 22
Population: Data are reported for evaluable participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | COB 80 mg + GDC 300 mg | COB 20 mg + GDC 200 mg | COB 40 mg + GDC 200 mg | COB 80 mg + GDC 200 mg | COB 80 mg + GDC 400 mg | COB 100 mg + GDC 200 mg
Number analyzed (Participants) | 1 | 5 | 3 | 5 | 4 | 6
nanograms per milliliter (ng/mL)
  Day 1: number analyzed (Participants) | 0 | 5 | 3 | 5 | 4 | 6
  Day 1 |  | 41.8 (102.0) | 90.2 (60.9) | 392 (31.9) | 155 (52.5) | 384 (53.2)
  Steady State: number analyzed (Participants) | 1 | 2 | 1 | 3 | 1 | 2
  Steady State | 73.0 | 48.5 (121.0) | 204 | 399 (46.4) | 284 | 431 (63.3)

16. Secondary Outcome: Median Time to Maximum Serum Concentration (Tmax) for Cobimetinib
Time Frame: Up to Day 22
Population: Data are reported for evaluable participants.
Measure: Median (Full Range); unit: hours
Arm/Group | COB 80 mg + GDC 300 mg | COB 20 mg + GDC 200 mg | COB 40 mg + GDC 200 mg | COB 80 mg + GDC 200 mg | COB 80 mg + GDC 400 mg | COB 100 mg + GDC 200 mg
Number analyzed (Participants) | 1 | 5 | 3 | 5 | 4 | 6
hours
  Day 1: number analyzed (Participants) | 0 | 5 | 3 | 5 | 4 | 6
  Day 1 |  | 2.00 [2.00 to 4.00] | 2.00 [1.00 to 3.00] | 2.00 [1.00 to 3.00] | 4.00 [2.00 to 6.00] | 2.00 [1.00 to 3.00]
  Steady State: number analyzed (Participants) | 1 | 2 | 1 | 3 | 1 | 2
  Steady State | 1.00 | 1.50 [1.00 to 2.00] | 24.0 | 1.00 [0.500 to 2.00] | 2.00 | 2.00 [2.00 to 2.00]

17. Secondary Outcome: Total Exposure (AUC From Time 0 to 24 Hour After Dose) for GDC-0994
Description: Data are reported for evaluable participants.
Time Frame: 0 to 24 hours post-dose (Up to Day 22)
Population: Data are reported for evaluable participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr x microM
Arm/Group | COB 80 mg + GDC 300 mg | COB 20 mg + GDC 200 mg | COB 40 mg + GDC 200 mg | COB 80 mg + GDC 200 mg | COB 80 mg + GDC 400 mg | COB 100 mg + GDC 200 mg
Number analyzed (Participants) | 1 | 5 | 3 | 5 | 4 | 6
hr x microM
  Day 1: number analyzed (Participants) | 0 | 5 | 3 | 5 | 4 | 6
  Day 1 |  | 37.0 (45.9) | 32.9 (55.4) | 27.9 (93.8) | 37.8 (37.5) | 37.7 (81.0)
  Steady State: number analyzed (Participants) | 1 | 2 | 1 | 3 | 1 | 1
  Steady State | 48.3 | 23.5 (73.4) | 24.1 | 33.3 (66.4) | 37.2 | 34.0

18. Secondary Outcome: Total Exposure (AUC From Time 0 to 24 Hour After Dose) for Cobimetinib
Time Frame: 0 to 24 hours post-dose (Up to Day 22)
Population: Data are reported for evaluable participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng x hr/mL
Arm/Group | COB 80 mg + GDC 300 mg | COB 20 mg + GDC 200 mg | COB 40 mg + GDC 200 mg | COB 80 mg + GDC 200 mg | COB 80 mg + GDC 400 mg | COB 100 mg + GDC 200 mg
Number analyzed (Participants) | 1 | 5 | 3 | 5 | 4 | 6
ng x hr/mL
  Day 1: number analyzed (Participants) | 0 | 5 | 3 | 5 | 4 | 6
  Day 1 |  | 501 (121.0) | 1020 (33.9) | 4420 (25.5) | 2460 (50.9) | 4060 (74.3)
  Steady State: number analyzed (Participants) | 1 | 2 | 1 | 3 | 1 | 1
  Steady State | 908 | 508 (255.0) | 2460 | 4320 (37.4) | 3410 | 4070

19. Secondary Outcome: Mean Accumulation Ratio
Time Frame: Pre-dose Day 1 Cycle 1, 2, 3, Day 18, 21 Cycle 1; post-dose 0.5, 1, 2, 3, 4, 6 hours Day 1, 18, 21 Cycle 1; Day 2, 15, 19, 22, Cycle 1
Population: Data for this measure were not collected.
Arm/Group | Not Assigned | COB 20 mg + GDC 200 mg | COB 40 mg + GDC 200 mg | COB 80 mg + GDC 200 mg | COB 80 mg + GDC 400 mg | COB 100 mg + GDC 200 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Mean Terminal Half-life (t1/2)
Time Frame: Up to day 22 of study
Population: Data for this measure were not collected.
Arm/Group | Not Assigned | COB 20 mg + GDC 200 mg | COB 40 mg + GDC 200 mg | COB 80 mg + GDC 200 mg | COB 80 mg + GDC 400 mg | COB 100 mg + GDC 200 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: Change From Baseline in Fluorodeoxyglucose Positron Emission Tomography (FDG-PET)
Time Frame: Baseline, Day 15
Population: Data for this measure were not collected.
Arm/Group | Not Assigned | COB 20 mg + GDC 200 mg | COB 40 mg + GDC 200 mg | COB 80 mg + GDC 200 mg | COB 80 mg + GDC 400 mg | COB 100 mg + GDC 200 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Change From Baseline in Tumor Tissue Biomarkers
Time Frame: Up to 15 months
Population: Data for this measure were not collected.
Arm/Group | Not Assigned | COB 20 mg + GDC 200 mg | COB 40 mg + GDC 200 mg | COB 80 mg + GDC 200 mg | COB 80 mg + GDC 400 mg | COB 100 mg + GDC 200 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 15 months
Arm/Group | Not Assigned | COB 20 mg + GDC 200 mg | COB 40 mg + GDC 200 mg | COB 80 mg + GDC 200 mg | COB 80 mg + GDC 400 mg | COB 100 mg + GDC 200 mg
Serious Adverse Events (participants affected / at risk) | 1/1 | 2/5 | 2/3 | 3/5 | 2/4 | 4/6
Other Adverse Events (participants affected / at risk) | 1/1 | 5/5 | 3/3 | 5/5 | 4/4 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Not Assigned (N=1) | COB 20 mg + GDC 200 mg (N=5) | COB 40 mg + GDC 200 mg (N=3) | COB 80 mg + GDC 200 mg (N=5) | COB 80 mg + GDC 400 mg (N=4) | COB 100 mg + GDC 200 mg (N=6)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTRIC ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHOLANGITIS INFECTIVE (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
KLEBSIELLA BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA VIRAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DISEASE PROGRESSION (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GAIT DISTURBANCE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Not Assigned (N=1) | COB 20 mg + GDC 200 mg (N=5) | COB 40 mg + GDC 200 mg (N=3) | COB 80 mg + GDC 200 mg (N=5) | COB 80 mg + GDC 400 mg (N=4) | COB 100 mg + GDC 200 mg (N=6)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 2 (3)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SINUS BRADYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SINUS TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DYSACUSIS (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DETACHMENT OF RETINAL PIGMENT EPITHELIUM (Eye disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
EYELID OEDEMA (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PERIORBITAL OEDEMA (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
PHOTOPHOBIA (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VISION BLURRED (Eye disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
VISUAL IMPAIRMENT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VITREOUS FLOATERS (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (3)
ASCITES (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
COLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 4 (5) | 2 (2) | 5 (10) | 4 (4) | 4 (8)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (2) | 5 (5) | 2 (2) | 4 (5) | 3 (3) | 2 (3)
SALIVARY GLAND ENLARGEMENT (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 3 (4) | 1 (1) | 5 (6) | 3 (4) | 3 (4)
ASTHENIA (General disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
CHILLS (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
FACE OEDEMA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
FATIGUE (General disorders) | 0 (0) | 4 (4) | 1 (1) | 2 (4) | 2 (5) | 3 (4)
GENERALISED OEDEMA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
LOCALISED OEDEMA (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 2 (3) | 1 (3) | 2 (2) | 1 (1) | 0 (0)
PERIPHERAL SWELLING (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ATYPICAL PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CANDIDA INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (9)
BLOOD ALBUMIN DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 2 (4)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BLOOD LACTIC ACID INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BLOOD UREA INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EJECTION FRACTION DECREASED (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
PROTEIN TOTAL DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TROPONIN INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
WEIGHT DECREASED (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 2 (2)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 2 (3) | 3 (3) | 2 (2) | 1 (1)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (2)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (2) | 1 (1) | 1 (1)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (2) | 0 (0) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
MALNUTRITION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ATAXIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BURNING SENSATION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LETHARGY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
SOMNOLENCE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VISUAL FIELD DEFECT (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DELIRIUM (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DYSURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ALVEOLAR LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TONSILLAR HYPERTROPHY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (3) | 2 (3) | 1 (1) | 4 (6) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
RASH MACULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SWELLING FACE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.